CLINICAL TRIAL: NCT04589897
Title: A Pilot Study Investigating the Effects of a Manuka Honey Sinus Rinse on Sino-nasal Outcome Test Scores in Cystic Fibrosis Patients
Brief Title: Manuka Honey Sinus Rinse Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: University Hospital of Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: JMR1075-100
Record Dates: First submitted 2020-09-24; First posted 2020-10-19 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2021-10

CONDITIONS: Cystic Fibrosis; Infection, Bacterial
MeSH Terms: conditions — Cystic Fibrosis; Bacterial Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Manuka honey sinus rinse
  Interventions: Device: Manuka honey sinus rinse
- Standard (Active Comparator): Standard sinus rinse
  Interventions: Device: Standard sinus rinse

INTERVENTIONS:
Device: Manuka honey sinus rinse — Will follow a modified NHS nasal rinse protocol with the addition of manuka honey
  Arms: Experimental
Device: Standard sinus rinse — will follow the standard NHS nasal rinse protocol
  Arms: Standard

SUMMARY:
A trial investigating the effect of a sinus rinse in people with CF

DETAILED DESCRIPTION:
People with with CF often have bacterial infection in their air ways. There is great interest in the different types of bacteria found within these infections.

This clinical trial looks at whether a novel sinus rinse device (that incorporates manuka honey) could help clear infection or reduce the amount and/or types of bacteria found within the upper airway. This study assesses the changes in the Sino-Nasal Outcome Test (SNOT-22) scores along with any changes in quality of life, before and after the use of a sinus rinse device for 30 days.

In addition to this, the amount and types of bacteria found in nasal swabs, the sinus rinse solution, and sputum samples, before and after using the sinus rinse device will be investigated. Sputum samples will also be monitored for changes in composition before and after using the sinus rinse.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to give informed consent.
* The patient must be ≥ 18 years.
* The patient must have an established diagnosis of CF (one or more of the following) Sweat chloride >60mEq/L Presence of two CF causing mutations.
* The patient must have chronic symptoms of rhinosinusitis according to the criteria of the European Position Paper on Rhinosinusitis (appendix A).
* The patient scores greater ≥ 7 on their SNOT-22 questionnaire.

Exclusion Criteria:

* The patient has ever tested positive for the bacteria Mycobacterium tuberculosis.
* The patient is currently using a nasal rinse protocol.
* The patient has undergone sinus surgery within 6 months.
* The patient suffers from nasal bleeding.
* The patient is currently undergoing systemic antibiotic therapy for infective exacerbation.
* The patient is using overnight oxygen via nasal cannula.
* The patient is participating in another clinical trial or has done so within the last 30 days.
* The patient has a known allergy to bee products.
* The patient has an objection to the use of bee products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Sino-Nasal Outcome Test 22 (SNOT- 22) Score | Baseline and day 30 (+-7 days)
  Does the addition of manuka honey to the sinus rinse change the Sino Nasal Outcome Test (SNOT)-22 score of patients with cystic fibrosis? The SNOT-22 scale runs from 0 -110 and a higher score indicating worse symptoms

SECONDARY OUTCOMES:
Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Score | Baseline and day 30 (+-7 days)
  Does the addition of manuka honey to a sinus rinse change the CFQ-R score in patients with cystic fibrosis? The scale runs from 1-100 and a higher score indicates a better outcome
Bacterial type and number | Baseline and day 30 (+-7 days)
  Does the addition of manuka honey to a sinus rinse impact on the bacterial type/amount found in the nasal/paranasal cavities of patients with cystic fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Duckers, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- All Wales Adult Cystic Fibrosis Center, University Hospital Llandough, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial that underlie the results to be reported in an article after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Derived] Roberts AEL, Xanthe C, Hopkins AL, Bodger O, Lewis P, Mahenthiralingam E, Duckers J, Jenkins RE. A pilot study investigating the effects of a manuka honey sinus rinse compared to a standard sinus rinse on sino-nasal outcome test scores in cystic fibrosis patients. Pilot Feasibility Stud. 2022 Sep 24;8(1):216. doi: 10.1186/s40814-022-01175-0. PMID 36153609

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04589897/Prot_SAP_000.pdf